CLINICAL TRIAL: NCT03685604
Title: Polyvinylpyrrolidone (PVP) Iodine vs Chlorhexidine in Alcohol for Disinfection of the Surgical Site: a Cluster-randomized Multicenter Trial
Brief Title: PVP Iodine vs Chlorhexidine in Alcohol for Disinfection of the Surgical Site
Acronym: PICASSo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-00962; me17Widmer2
Record Dates: First submitted 2018-09-10; First posted 2018-09-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Surgical Site Infections
Keywords: chlorhexidine in alcoholic solution; PVP iodine in alcoholic solution; preoperative skin antisepsis
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: The intervention will be conducted as an open-label cluster-randomized cross-over multicenter trial with an allocation ratio of 1:1.
  The departments of surgery of the 3 study sites will be randomized center-wise in clusters by month to use CHX or PI. The products will be switched over according to the computer-generated randomization list.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cardiothoracic surgery - PI disinfection (Active Comparator)
  Interventions: Drug: PI Disinfection
- Cardiothoracic surgery - CHX disinfection (Active Comparator)
  Interventions: Drug: CHX disinfection
- Abdominal surgery - PI disinfection (Active Comparator)
  Interventions: Drug: PI Disinfection
- Abdominal surgery - CHX disinfection (Active Comparator)
  Interventions: Drug: CHX disinfection

INTERVENTIONS:
Drug: CHX disinfection — CHX (Softasept® Chlorhexidine solution 2% coloured, from B. Braun Medical AG) is applied three times on the patient's skin with the use of swabs. The cumulative residence time is a minimum of 3 minutes. The application is performed according to standard procedures of the participating centers and according to manufacturer's recommendations
  Arms: Abdominal surgery - CHX disinfection; Cardiothoracic surgery - CHX disinfection
Drug: PI Disinfection — PI (Braunoderm® from B.Braun or Betaseptic® from Mundipharma) is applied prior to surgery on the patient's skin with the use of swabs. The product is applied three times. The cumulative residence time is a minimum of 3 minutes. The application is performed according to standard procedures of the participating centers and according to manufacturer's recommendations
  Arms: Abdominal surgery - PI disinfection; Cardiothoracic surgery - PI disinfection

SUMMARY:
Prospective cluster-randomized multicenter cross-over trial to prove non-inferiority of PI compared to CHX in preoperative skin antisepsis

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are the most common nosocomial infections in surgical patients causing significant increases in morbidity, mortality, and health care costs. As they are usually caused by components of the normal skin flora, disinfection of the surgical site with an antiseptic skin preparation is standard practice prior to any surgical intervention. The most commonly used disinfectants are either chlorhexidine in alcoholic solution (CHX) or PVP iodine in alcoholic solution (PI) This prospective cluster-randomized multicenter cross-over trial is to prove non-inferiority of PI compared to CHX in preoperative skin antisepsis in abdominal and cardiothoracic surgery in regard of SSIs.

ELIGIBILITY:
Inclusion Criteria:

- undergoing cardiac or certain types of abdominal surgery (colorectal surgery, cholecystectomy, herniotomy, appendectomy and bariatric surgery) which are routinely followed up by the study Centers during the study period

Exclusion Criteria:

* contraindication to the use of either one of the compounds ( CHX: intolerance to any of the compounds of the preparation, application on cornea, wounds or mucosal Membrane. PI: hyperthyroid disease, intolerance to any of the compounds, iodine allergy, 2 weeks prior to radio- iodine treatment, Dermatitis herpetiformis Duhring, application on cornea, wounds or mucosal membranes)
* Emergency surgical Intervention
* Patients refusing General consent for use of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3321 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infections (SSIs) | occurrence of surgical site infections is evaluated at three time points: at time of dismissal from the hospital (approx. 1 week after surgical intervention); 30 days after abdominal and cardiac surgery; 1 year for cardiac surgery
  Comparison of SSI rates between the two groups using standard chi-square test. Presence of SSIs for abdominal and cardiac surgeries as defined by Swiss society of hospital epidemiologists (Swissnoso) according to National Healthcare Safety Network (NHSN) criteria. Analysis will be performed using the final SSI rate (30 days for abdominal, 30 days/1 year for cardiac surgery) and according to the different types of infections. Infection ratio will be calculated as crude ratio as well as adapted to the National Nosocomial Infections Surveillance System (NNIS) score. The method of aggregation for the combined SSI rate for both types of surgery together will be a weighted average based on the proportion of SSIs from each surgery type. The measure includes no scale.

SECONDARY OUTCOMES:
Type of SSI: superficial, deep, organ-space | three time points: at time of dismissal from the hospital (approx. 1 week after surgical intervention); 30 days after abdominal and cardiac surgery; 1 year for cardiac surgery
  Type of SSI: superficial, deep, organ-space; DEFINITIONS OF SSI: For surveillance classification purposes, SSIs are divided into incisional SSIs and organ/space SSIs. Incisional SSIs are further classified into those involving only the skin and subcutaneous tissue (called superficial incisional SSIs) and those involving deep soft tissues of the incision (called deep incisional SSIs (e.g., fascial and muscle layers)). Organ/space SSIs involve any part of the anatomy (e.g., organs or spaces), other than the incision, opened or manipulated during the operative procedure.
Body Mass Index (BMI) | day of surgery
  Subgroup analysis stratified by patient factors (i.e. BMI). Weight and height will be combined to report BMI in kg/m^2).
Change in hemoglobin (g/l) | day of surgery
  Subgroup analysis stratified by laboratory parameters: hemoglobin (g/l)
Mortality | in-hospital (approx. 1 week from surgical intervention) and 30 day for abdominal surgery; in-hospital (approx. 1 week from surgical intervention), 30 day and 365 day for cardiac surgery
  death rate
Timing of antimicrobial prophylaxis | day of surgery
  Timing of antimicrobial prophylaxis (antibiotic, dose,time of application)
Duration of surgery | time from start to stop of surgical intervention
  Duration of surgery
Wound contamination -class according to Centers for Disease Control and Prevention(CDC) | three time points: at time of dismissal from the hospital (approx. 1 week after surgical intervention); 30 days after abdominal and cardiac surgery; 1 year for cardiac surgery
  Wound contamination -class according to Centers for Disease Control and Prevention(CDC)
American Society of Anesthesiologists (ASA) -score | day of surgery
  ASA physical status classification system is a system for assessing the fitness of patients before surgery. These are:
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  6. A declared brain-dead person whose organs are being removed for donor purposes.
Change in creatinine (ymol/l) | in- hospital stay (approx. 1 week from surgical intervention)
  Subgroup analysis stratified by laboratory parameters: creatinine (ymol/l)
Change in leukocytes (x10^9/l) | in- hospital stay (approx. 1 week from surgical intervention)
  Subgroup analysis stratified by laboratory parameters: leukocytes (x10^9/l)
Change in concentration for C reactive Protein (CRP) (mg/l) | in- hospital stay (approx. 1 week from surgical intervention)
  Subgroup analysis stratified by laboratory parameters: CRP (mg/l)
National Nosocomial Infections Surveillance System (NNIS) index | in- hospital stay (approx. 1 week from surgical intervention)
  NNIS index takes into account 3 risk factors, and each is awarded 1 point: contaminated or dirty-infected surgical wound, American Society of Anesthesiology (ASA) score greater than 2 and surgery duration longer than T (where T is defined as the 75th percentile of the average time for a surgical procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Widmer, Prof. Dr. MD, Principal Investigator — University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology, Basel
  - University Hospital of Bern; Division of Infectious Diseases and Hospital Epidemiology, Bern
  - University Hospital Zurich, Division of Infectious Diseases and Hospital Epidemiology, Zurich

REFERENCES:
- [Derived] Widmer AF, Atkinson A, Kuster SP, Wolfensberger A, Klimke S, Sommerstein R, Eckstein FS, Schoenhoff F, Beldi G, Gutschow CA, Marschall J, Schweiger A, Jent P. Povidone Iodine vs Chlorhexidine Gluconate in Alcohol for Preoperative Skin Antisepsis: A Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):541-549. doi: 10.1001/jama.2024.8531. PMID 38884982